CLINICAL TRIAL: NCT05108311
Title: Effectiveness of a Novel Protocol for Glenohumeral Internal Rotation Deficit in General Population With Shoulder Pain
Acronym: GIRDTREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEU-024
Record Dates: First submitted 2021-10-22; First posted 2021-11-04 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2021-10

CONDITIONS: Shoulder Pain; Glenohumeral Internal Rotation Deficit
Keywords: general population.; Manual therapy; Therapeutic Exercise
MeSH Terms: conditions — Shoulder Pain | interventions — Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The Treatment sequence including joint Manual therapy techniques and soft tissue release techniques is proposed.
  Interventions: Other: Manual therapy and therapeutic exercise

INTERVENTIONS:
Other: Manual therapy and therapeutic exercise — 1. Gliding over the deltoid superficial fascia.
  2. Anterior-Posterior mobilization of the clavicle.
  3. myofascial release of the shoulder joint complex techniques.
  4. Myofascial release external rotation with glenohumeral decoaptation will be carry out in prone position facility the triangular space, quadrangular space and triceps hiatus.
  5. anterior and posterior, superior and inferior glenohumeral inferior glide mobilization in adduction will perform in a prone position to facilitate glenohumeral re centration.
  6. scapular musculature myofascial release including mobilization with a scapulothoracic joint decoaptation, and angular of the scapula.
  7. Supine mobilization of the posterior capsule in 90º shoulder flexion and the adduction.
  Finally the patient will be instructed to adapt the daily active biological stimulus at home to maximize the benefits of the manual therapy

SUMMARY:
Shoulder pain is one of the most common joint problems and disabling complaint in general population., but there is a lack of evidence about the relation between shoulder pain and glenohumeral internal rotation deficit (GIRD) in general population.

This study aimed to determine if the novel proposal for treatment of GIRD could be effectiveness and gain further evidence in the Range of Motion an Pain.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain

Exclusion Criteria:

* Patient under 18 years old,
* Pain in both shoulders
* Joint prosthesis in at least one of the two shoulders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
glenohumeral internal rotation | Baseline
  measure in supine position on a physiotherapy bench. The shoulder will held at 90° abduction with 90° flexion in the elbow.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Jácome López, PT, Principal Investigator — Clínica Universidad de Navarra
Locations (1):
- San Pablo CEU University, Boadilla del Monte, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided